CLINICAL TRIAL: NCT03349164
Title: Local Registry of Patients With Chronic Thromboembolic Pulmonary Hypertension in Novosibirsk Region
Brief Title: Registry of Patients With Chronic Thromboembolic Pulmonary Hypertension in Novosibirsk Region
Acronym: NCTEPHR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Novosibirsk Scientific Research Institute for Circulatory Pathology (Other)
Responsible Party: Sponsor
Other Study IDs: NCTEPHR
Record Dates: First submitted 2017-11-12; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: acute PE survivors — Patients from this group will be assessed by cardiologist, echocardiography and VQ scanning

SUMMARY:
There will be assessment of patients after acute pulmonary embolism for the development of CTEPH

DETAILED DESCRIPTION:
There will be assessment of patients after acute pulmonary embolism for the development of CTEPH.

There will be analysis of case histories of 40 patients with acute pulmonary embolism. All this patients will be clinically assessed by local cardiologist. Also echocardiography, lung VQ scans (perfusion and ventilation) will be performed.

Patients with chronic thromboembolic pulmonary hypertension will be assessed by local team experienced in CTEPH treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients who had episodes of acute pulmonary embolism
* 3-4 months of anticoagulation treatment after acute pulmonary embolism
* informed consent

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are survivors after acute PE. Than they should intake anticoagulation treatment at least 3-4 month. Then they will be assessed clinically by local cardiologists, echocardiography and VQ scan will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2018-03-10 (Estimated)

PRIMARY OUTCOMES:
clinical presentation of chronic thromboembolic pulmonary hypertension | 3-4 month after acute pulmonary embolism
  presence of dyspnea after acute pulmonary embolism will be the sign of clinical symptomatic patients. Dyspnea will be assessed with Borg scale
clinical presentation of chronic thromboembolic pulmonary hypertension | 3-4 month after acute pulmonary embolism
  clinical assessment of physical capacity of patient with 6 minute walking distance test and NYHA functional class

SECONDARY OUTCOMES:
presence of pulmonary hypertension - mean pulmonary artery pressure > 25 mm Hg according to echocardiography | 3-4 month after acute pulmonary embolism
  presence of pulmonary hypertension - mean pulmonary artery pressure > 25 mm Hg according to echocardiography
presence of perfusion deficit in pulmonary artery according to VQ scan | 3-4 month after acute pulmonary embolism
  presence of perfusion deficit in pulmonary artery according to VQ scan

CONTACTS AND LOCATIONS:
Locations (1):
- Novosibirsk research institute of circulation pathology, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided